CLINICAL TRIAL: NCT03219190
Title: A High School Program for Preventing Prescription Drug Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Promotion Associates, Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Williams, Senior Research Scientist, National Health Promotion Associates, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R44DA04327301
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prescription Drug Abuse; Substance Abuse; Substance Use (Drugs, Alcohol)
Keywords: Adolescence; Prescription Drug Misuse; Prevention; Hybrid; E-learning; Cigarette Smoking; Alcohol Use; Life Skills
MeSH Terms: conditions — Substance-Related Disorders; Prescription Drug Misuse; Cigarette Smoking; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LST High School Hybrid (Experimental): Provided with the prevention program, consisting of e-learning modules and classroom sessions.
  Interventions: Behavioral: LST High School Hybrid
- Treatment as Usual (Control) (No Intervention): Standard health education

INTERVENTIONS:
Behavioral: LST High School Hybrid — The preventive intervention for high school PDM will: (1) utilize both online e-learning modules and interactive classroom sessions to address PDM and concurrent alcohol/drug abuse; (2) positively change social norms surrounding PDM and alcohol/drug abuse; (3) change positive expectancies about the benefits of PDM; (4) discourage diversion of prescription medication; (5) enhance protective factors by building social, self-regulation, and relationship skills through interactive learning and behavioral rehearsal scenarios; and (6) include online booster sessions.
  Arms: LST High School Hybrid

SUMMARY:
This project will develop and evaluate a program to prevent prescription drug misuse in high school students

DETAILED DESCRIPTION:
This Fast-Track SBIR project is designed to address the critical need for an effective primary prevention approach for prescription misuse (PDM), an urgent public health crisis in the United States. The project involves developing and testing an innovative new approach to the primary prevention of PDM among high school students utilizing e-learning and small group facilitator-led intervention modalities. The intervention is an adaptation of the evidence-based substance abuse prevention approach called Life Skills Training (LST). The adapted intervention will address the relationship between PDM and alcohol, tobacco and other drug (ATOD) use and abuse; positively change social norms surrounding ATOD and PDM; discourage diversion of prescription medications; enhance protective factors by building social and self-regulation skills through interactive learning and behavioral rehearsal scenarios.

Administrative Correction: This record was updated post-study to rectify administrative errors in the original registration and to reflect operational changes necessitated by the COVID-19 pandemic.

Correction of Secondary Outcomes: The Secondary Outcomes section has been corrected to include variables that were specified in several sections of the original registration and collected during the trial, but were inadvertently omitted from the "Outcome Measures" field in the initial registration. These include: alcohol use, tobacco use, marijuana use, inhalant use, perceived risk of prescription sedative, painkiller, and stimulant misuse, and life skills (self-regulation, communication, media resistance, anxiety management, refusal skills).

Update on Study Duration and Follow-up: The COVID-19 pandemic caused significant delays in study implementation and data collection. Although the original protocol specified 12- and 24-month follow-ups, the 24-month assessment was canceled because the study delays extended the timeline beyond the NIH/NIDA performance period. Additionally, widespread school closures and access restrictions resulted in high attrition at the 12-month time point, rendering those data insufficient for meaningful analysis. Consequently, the study analysis focuses exclusively on the immediate post-intervention timeframe.

Clarification on Terminology: Although our original grant application and ClinicalTrials.gov registration used the term Prescription Drug Abuse (PDA), we have adopted the more contemporary term Prescription Drug Misuse (PDM) to align with current best practices. PDM is defined here as the use of prescription drugs without a doctor's prescription.

ELIGIBILITY:
Correction of Minimum and Maximum Ages: The correct minimum and maximum age range for the study population is ages 14-18.

Inclusion Criteria:

* High school aged-youth

Exclusion Criteria:

* Significant cognitive impairment or severe learning disabilities, as screened by field staff at participating sites

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1804 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Prescription Drug Misuse (i.e., prescription drug use without a doctor's prescription) | Pre-test and post-test assessment (approx 2-4 weeks post-intervention)
  This measure includes prescription drug misuse of sedatives, painkillers, and stimulants.
  Frequency of sedative, painkiller, and stimulant use without a doctor's prescription; measured on a 9-point scale, including Never (1), A few times but NOT in the past year (2), A few times a year (3), Once a month (4), A few times a month (5), Once a week (6), A few times a week (7), Once a day (8), More than once a day (9)

SECONDARY OUTCOMES:
Alcohol Use | Pre-test and post-test assessment (approx 2-4 weeks post-intervention)
  This measure includes alcohol use and alcohol intoxication. Frequency of alcohol use and alcohol intoxication; measured on a 9-point scale, including Never (1), A few times but NOT in the past year (2), A few times a year (3), Once a month (4), A few times a month (5), Once a week (6), A few times a week (7), Once a day (8), More than once a day (9)
Tobacco Use | Pre-test and post-test assessment (approx 2-4 weeks post-intervention)
  This measure includes tobacco use. Frequency of cigarette/tobacco use; measured on a 9-point scale, including Never (1), A few times but NOT in the past year (2), A few times a year (3), Once a month (4), A few times a month (5), Once a week (6), A few times a week (7), Once a day (8), More than once a day (9)"
Marijuana Use | Pre-test and post-test assessment (approx 2-4 weeks post-intervention)
  This measure includes marijuana use. Frequency of marijuana use; measured on a 9-point scale, including Never (1), A few times but NOT in the past year (2), A few times a year (3), Once a month (4), A few times a month (5), Once a week (6), A few times a week (7), Once a day (8), More than once a day (9)"
Inhalant Use | Pre-test and post-test assessment (approx 2-4 weeks post-intervention)
  This measure includes inhalant use; measured on a 9-point scale, including Never (1), A few times but NOT in the past year (2), A few times a year (3), Once a month (4), A few times a month (5), Once a week (6), A few times a week (7), Once a day (8), More than once a day (9)"
Substance Use Intentions | Pre-test and post-test assessment (approx 2-4 weeks post-intervention)
  This measure includes intentions to use substances: Intentions to use alcohol, get drunk, use tobacco, marijuana, and inhalants within the next year; measured on a 5-point scale from "Definitely Not" to "Definitely Will"
Perceived Risk of Prescription Drug Misuse | Pre-test and post-test assessment (approx 2-4 weeks post-intervention)
  This measure includes perceived risk of harm associated with using prescription sedatives, painkillers, and stimulants when prescribed for someone else, measured on a 4-point scale from "No Risk" to "Great Risk;" also option for "Can't say, drug unfamiliar."

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Williams, PhD, MPH, Principal Investigator — National Health Promotion Associates, Inc.
Locations (1):
- National Health Promotion Associates, Inc., White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Retraction of "Preventing tobacco and alcohol use among high school students through a hybrid online and in-class intervention: A randomized controlled trial," by Williams et al. (2025). Psychol Addict Behav. 2026 Feb;40(1):125. doi: 10.1037/adb0001131. PMID 41627337